CLINICAL TRIAL: NCT04464265
Title: Magnetic Resonance Imaging of the Effect of Music Listening on Brain Activity Under Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Anthony G Hudetz, Professor of Anesthesiology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00176300; R01GM103894 (NIH)
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Healthy
Keywords: Music; Propofol
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Functional Magnetic Resonance Imaging (Experimental): While music is played Noninvasive functional magnetic resonance (fMRI) imaging will be performed at the University of Michigan Health System, University Hospital, Department of Radiology.
  The fMRI is done under anesthesia using propofol. The researchers will manually control the infusion of propofol to achieve target effect-site concentrations of 1.2, 1.6, 2.0, and 2.4 μg/ml in a stepwise fashion.
  Interventions: Other: Functional Magnetic Resonance Imaging (fMRI)

INTERVENTIONS:
Other: Functional Magnetic Resonance Imaging (fMRI) — Propofol will be administered by intravenous infusion. All anesthesia equipment, supplies, and drugs will be provided by anesthesiologists from the University of Michigan Health System. The researchers will manually control the infusion of propofol to achieve target effect-site concentrations which will be maintained for 4 minutes each.
  Four types of music, including Jazz, Rock, Pop and Country, will be presented in a pseudo-randomized order. During the behavioral test period, participants will be asked to squeeze an Magnetic Resonance Imaging (MRI) compatible grip dynamometer (a rubber ball) for every 10-second periods (96 cycles in total). The beginning of each cycle will be cued with the spoken word "squeeze".
  Other Names: Diprivan

SUMMARY:
This study is to better understand the systems-level neuronal mechanisms by which general anesthetics produce loss of consciousness.The researchers believe that anesthetics suppress consciousness by disrupting the functioning of large-scale brain networks that support information integration in the brain.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist physical status of 1 (ASA-1), Healthy, non-smoking, no or minimal alcohol use
* Right-handed
* Body mass index (BMI) of less than 30
* English speakers

Exclusion Criteria:

* Medical contraindication to Magnetic Resonance Imaging (MRI) scanning
* Unable to undergo MRI scanning because of possible pregnancy
* BMI over 30
* Tattoos in the head or neck region
* Unwilling to abstain from alcohol for 24 hours prior to dosing

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Hudetz, PhD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Functional Magnetic Resonance Imaging: While music is played Noninvasive functional magnetic resonance (fMRI) imaging will be performed at the University of Michigan Health System, University Hospital, Department of Radiology.
  The fMRI is done under anesthesia using propofol. The researchers will manually control the infusion of propofol to achieve target effect-site concentrations of 1.2, 1.6, 2.0, and 2.4 μg/ml in a stepwise fashion.
  Functional Magnetic Resonance Imaging (fMRI): Propofol will be administered by intravenous infusion. All anesthesia equipment, supplies, and drugs will be provided by anesthesiologists from the University of Michigan Health System. The researchers will manually control the infusion of propofol to achieve target effect-site concentrations which will be maintained for 4 minutes each.
  Four types of music, including Jazz, Rock, Pop and Country, will be presented in a pseudo-randomized order. During the behavioral test period, participants will be asked to squeeze an Magnetic Resonance Imaging (MRI) compatible grip dynamometer (a rubber ball) for every 10-second periods (96 cycles in total). The beginning of each cycle will be cued with the spoken word "squeeze".
Period: Overall Study
Arm/Group | Functional Magnetic Resonance Imaging
Started | 32
Completed | 30
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: While 47 participants were consented, 15 dropped out prior to receiving the intervention.
Arm/Group | Functional Magnetic Resonance Imaging
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (0.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Blood Oxygen Level Dependent (BOLD) Response to Sensory Stimuli During Sedation
Description: Music evoked activity was quantified by measurements of the fMRI BOLD signal. Neural response to a natural auditory stimulus, music, was assessed during both conscious and anesthetized states. Measurements were taken at baseline (30 minutes) and during anesthesia (60 minutes).
Time Frame: 60 minutes
Population: Reason of excluding 3 subjects: there were large head motions during fMRI so that the results were not analyzed or pooled in the whole study group. Two additional subjects were excluded, as they withdrew due to physician discretion.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Functional Magnetic Resonance Imaging
Number analyzed (Participants) | 27
arbitrary units
  Baseline (at 30 minutes) | 0.04 (0.02)
  During Anesthesia (at 60 Minutes) | 0.01 (0.01)
Statistical Analysis 1: Comparison: Functional Magnetic Resonance Imaging; The null hypothesis is no difference in BOLD response between sedated state and baseline. For an fMRI study of cognitive function, Desmond and Glover (J. Neurosci. Methods., 2002) reported that about 25 subjects are necessary to achieve 80% power for a 0.5% increase of activity. We analyzed 27 subjects that fulfilled the suggested optimal group size for reliable statistics in functional MRI studies (also see Thirion et al., Neuroimage, 2007); Test type: Other — Our study adopted a within-subject design, which is not a randomized controlled trial (RCT). The P-value below indicates if propofol administration has a statistically significant impact on the brain activity in response to sensory stimuli; p < 0.001, t-test, 2 sided — The threshold for statistical significance was p=0.05. The p-value was not adjusted for multiple comparisons, as only one comparison was performed; Mean Difference (Net) = -3, Standard Deviation 2 — Difference = BOLD Response During Sedation - BOLD Response During Baseline

2. Secondary Outcome: Average Squeeze Pressure Over 60 Minutes
Description: Measurement of force of participants' hand squeezing on a rubber ball in response to instructions. This will be measured in millimeters of mercury (mmHg) of air pressure during squeezing the rubber ball. Measurements are provided for the 30-minute means based on measurements taken every 10 seconds for 30 minutes prior to intervention (baseline) and every 10 seconds for 30 minutes during intervention (intervention), using BIOPAC (https://www.biopac.com) MP160 system with AcqKnowledge software (V5.0).
Time Frame: 60 minutes
Population: Two subjects were excluded, as they withdrew due to physician discretion.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Functional Magnetic Resonance Imaging
Number analyzed (Participants) | 30
mmHg
  Baseline (at 30 minutes) | 11.64 (4.01)
  Intervention (at 60 minutes) | 8.92 (4.11)
Statistical Analysis 1: Comparison: Functional Magnetic Resonance Imaging; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -2.72, Standard Deviation 3.17 — Difference = Squeeze Pressure During Sedation - Squeeze Pressure During Baseline

ADVERSE EVENTS:
Time Frame: 24 hours after drug adminstration
Arm/Group | Functional Magnetic Resonance Imaging
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Functional Magnetic Resonance Imaging (N=30)
Near syncope (Surgical and medical procedures) | 1 (1) — Participant experienced near syncope during IV insertion
Paresthesia (Surgical and medical procedures) | 1 (1) — Participant experienced paresthesia near IV insertion site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT04464265/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT04464265/ICF_000.pdf